CLINICAL TRIAL: NCT04852666
Title: Comparative Effectiveness of Biologics or Small Molecule Therapies After Failure of Anti-TNF Treatment in Patients With Crohn's Disease and Ulcerative Colitis
Brief Title: Comparative Effectiveness of Biologics or Small Molecule Therapies in Inflammatory Bowel Disease (IBD)
Acronym: COMPARE
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Crohn's and Colitis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 19-0273; PaCR-2017C2-8172-IC (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Results first posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-01

CONDITIONS: Crohn's Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Crohn's Disease (Vedolizumab): Participants with Crohn's disease (CD) who reported taking vedolizumab.
- Crohn's Disease (Ustekinumab): Participants with Crohn's disease (CD) who reported taking ustekinumab.
- Ulcerative Colitis (Vedolizumab): Participants with Ulcerative colitis (UC) who reported taking vedolizumab.
- Ulcerative Colitis (Tofacitinib): Participants with Ulcerative colitis (UC) who reported taking tofacitinib.

SUMMARY:
The purpose of this study is to assess effectiveness of vedolizumab versus ustekinumab in patients with Crohn's disease and vedolizumab versus tofacitinib in patients with ulcerative colitis, after non-response to anti-tumor necrosis factor (TNF) medications, using data from two existing cohorts.

DETAILED DESCRIPTION:
This study is a secondary analysis using data from participants in the IBD Partners and SPARC-IBD cohorts. Data received from IBD Partners consists of patient-reported outcomes gathered via online surveys (baseline and 6-month follow-ups). Data received from SPARC-IBD consists of patient-reported outcomes gathered via surveys (baseline and follow-ups) as well as data from clinical records.

ELIGIBILITY:
Inclusion Criteria:

* age greater than or equal to 18;
* diagnosis of CD or UC (as reported by participant for IBD Partners registry and/or physician for SPARC-IBD cohort);
* initiated vedolizumab or ustekinumab for CD, or initiated vedolizumab or tofacitinib for UC; treated with anti-TNF prior to vedolizumab/ustekinumab/tofacitinib.

Exclusion Criteria:

* less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population: participants in IBD Partners or SPARC cohort.
Sampling Method: Non-Probability Sample
Enrollment: 465 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kappelman, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - Crohn's & Colitis Foundation, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Crohn's Disease (Vedolizumab) | Crohn's Disease (Ustekinumab) | Ulcerative Colitis (Vedolizumab) | Ulcerative Colitis (Tofacitinib)
Started | 141 | 219 | 72 | 33
Completed | 141 | 219 | 72 | 33
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Crohn's Disease (Vedolizumab) | Crohn's Disease (Ustekinumab) | Ulcerative Colitis (Vedolizumab) | Ulcerative Colitis (Tofacitinib) | Total
Number analyzed (Participants) | 141 | 219 | 72 | 33 | 465
Age, Continuous [Median (Full Range); unit: years] | 44 [21 to 78] | 45 [18 to 79] | 42.5 [19 to 75] | 38 [19 to 74] | 42 [18 to 79]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 100 | 167 | 48 | 17 | 332
  Male | 41 | 52 | 20 | 14 | 127
  Data unavailable | 0 | 0 | 4 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 129 | 193 | 57 | 28 | 407
  Black or African American | 2 | 2 | 3 | 1 | 8
  Hispanic | 3 | 3 | 1 | 0 | 7
  Other or Unknown | 7 | 21 | 11 | 4 | 43

OUTCOME MEASURES:

1. Primary Outcome: PROMIS Measures of Pain Interference
Description: NIH Patient Reported Outcome Measurement Information System (PROMIS) measures of Pain Interference. PROMIS scores can range from 0 to 100; scales are calibrated using a T-score metric with a mean of 50 and standard deviation of 10. A higher score indicates more pain interference (poorer health).
Time Frame: Single assessment, performed as close to 6 months after medication initiation as possible (4-10 month window)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Crohn's Disease (Vedolizumab) | Crohn's Disease (Ustekinumab) | Ulcerative Colitis (Vedolizumab) | Ulcerative Colitis (Tofacitinib)
Number analyzed (Participants) | 141 | 219 | 72 | 33
T-score | 51.2 (10.17) | 51.6 (9.94) | 50.1 (10.2) | 48.2 (9.0)
Statistical Analysis 1: Comparison: Crohn's Disease (Vedolizumab) vs Crohn's Disease (Ustekinumab); Test type: Superiority; p = 0.751, t-test, 2 sided
Statistical Analysis 2: Comparison: Ulcerative Colitis (Vedolizumab) vs Ulcerative Colitis (Tofacitinib); Test type: Superiority; p = 0.372, t-test, 2 sided

2. Primary Outcome: PROMIS Measures of Fatigue
Description: NIH Patient Reported Outcome Measurement Information System (PROMIS) measures of Fatigue. PROMIS scores can range from 0 to 100; scales are calibrated using a T-score metric with a mean of 50 and standard deviation of 10. A higher score indicates more fatigue (poorer health).
Time Frame: Single assessment, performed as close to 6 months after medication initiation as possible (4-10 month window)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Crohn's Disease (Vedolizumab) | Crohn's Disease (Ustekinumab) | Ulcerative Colitis (Vedolizumab) | Ulcerative Colitis (Tofacitinib)
Number analyzed (Participants) | 141 | 219 | 72 | 33
T-score | 54.7 (11.73) | 54.4 (12.31) | 52.7 (11.8) | 50.6 (9.4)
Statistical Analysis 1: Comparison: Crohn's Disease (Vedolizumab) vs Crohn's Disease (Ustekinumab); Test type: Superiority; p = 0.778, t-test, 2 sided
Statistical Analysis 2: Comparison: Ulcerative Colitis (Vedolizumab) vs Ulcerative Colitis (Tofacitinib); Test type: Superiority; p = 0.357, t-test, 2 sided

3. Secondary Outcome: Number of Participants With Index Medication Persistence
Description: Medication persistence was defined as continuing index medication.
Time Frame: 4-10 months after medication initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease (Vedolizumab) | Crohn's Disease (Ustekinumab) | Ulcerative Colitis (Vedolizumab) | Ulcerative Colitis (Tofacitinib)
Number analyzed (Participants) | 141 | 219 | 72 | 33
Participants | 119 | 203 | 63 | 29
Statistical Analysis 1: Comparison: Crohn's Disease (Vedolizumab) vs Crohn's Disease (Ustekinumab); Test type: Superiority; p = 0.012, Chi-squared
Statistical Analysis 2: Comparison: Ulcerative Colitis (Vedolizumab) vs Ulcerative Colitis (Tofacitinib); Test type: Superiority; p = 0.956, Chi-squared

4. Secondary Outcome: Number of Participants Using Corticosteroids at Follow-Up
Description: Participants who reported using corticosteroids.
Time Frame: 4-10 months after medication initiation
Population: All available data are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease (Vedolizumab) | Crohn's Disease (Ustekinumab) | Ulcerative Colitis (Vedolizumab) | Ulcerative Colitis (Tofacitinib)
Number analyzed (Participants) | 141 | 219 | 71 | 30
Participants | 27 | 28 | 15 | 1
Statistical Analysis 1: Comparison: Crohn's Disease (Vedolizumab) vs Crohn's Disease (Ustekinumab); Test type: Superiority; p = 0.103, Chi-squared
Statistical Analysis 2: Comparison: Ulcerative Colitis (Vedolizumab) vs Ulcerative Colitis (Tofacitinib); Test type: Superiority; p = 0.025, Chi-squared

5. Secondary Outcome: Short Crohn's Disease Activity Index (sCDAI)
Description: Short Crohn's Disease Activity Index. This is a method to measure Crohn's disease patients' symptoms using only a questionnaire, which can be completed without an office visit or lab work. The variables included in the short CDAI are abdominal pain, stool frequency, and general well-being reported as a total score. The higher the score, the worse the disease activity. The sCDAI uses the same scale as the full CDAI with scores ranging from 0 to 600, such that scores,<150 define remission, 150 to 219 mild activity, 220 to 450 moderate activity, and greater than 450 severe activity.
Time Frame: Single assessment, performed as close to 6 months after medication initiation as possible (4-10 month window)
Population: This outcome applies only to those participants who have Crohn's disease.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crohn's Disease (Vedolizumab) | Crohn's Disease (Ustekinumab) | Ulcerative Colitis (Vedolizumab) | Ulcerative Colitis (Tofacitinib)
Number analyzed (Participants) | 141 | 219 | 0 | 0
score on a scale | 147 (89.6) | 144 (85.8) |  |
Statistical Analysis 1: Comparison: Crohn's Disease (Vedolizumab) vs Crohn's Disease (Ustekinumab); Test type: Superiority; p = 0.785, t-test, 2 sided

6. Secondary Outcome: Mayo Clinic Score
Description: The Mayo Clinic Score (MCS) asks 2 questions about (1) stool frequency and (2) rectal bleeding with an overall score range (0-6). Higher scores reflect more disease symptomatology.
Time Frame: Single assessment, performed as close to 6 months after medication initiation as possible (4-10 month window)
Population: This outcome applies only to those participants who have ulcerative colitis. All available data are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crohn's Disease (Vedolizumab) | Crohn's Disease (Ustekinumab) | Ulcerative Colitis (Vedolizumab) | Ulcerative Colitis (Tofacitinib)
Number analyzed (Participants) | 0 | 0 | 69 | 30
score on a scale |  |  | 1.7 (1.8) | 1.2 (1.5)
Statistical Analysis 1: Comparison: Ulcerative Colitis (Vedolizumab) vs Ulcerative Colitis (Tofacitinib); Test type: Superiority; p = 0.200, t-test, 2 sided

7. Secondary Outcome: PROMIS Social Satisfaction Score
Description: NIH Patient Reported Outcome Measurement Information System (PROMIS) measures of social satisfaction. PROMIS scores can range from 0 to 100; scales are calibrated using a T-score metric with a mean of 50 and standard deviation of 10. A higher score for social satisfaction indicates better health.
Time Frame: Single assessment, performed as close to 6 months after medication initiation as possible (4-10 month window)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Crohn's Disease (Vedolizumab) | Crohn's Disease (Ustekinumab) | Ulcerative Colitis (Vedolizumab) | Ulcerative Colitis (Tofacitinib)
Number analyzed (Participants) | 141 | 219 | 72 | 33
T-score | 49.1 (10.59) | 49.3 (10.06) | 47.5 (11.0) | 50.4 (10.6)
Statistical Analysis 1: Comparison: Crohn's Disease (Vedolizumab) vs Crohn's Disease (Ustekinumab); Test type: Superiority; p = 0.887, t-test, 2 sided
Statistical Analysis 2: Comparison: Ulcerative Colitis (Vedolizumab) vs Ulcerative Colitis (Tofacitinib); Test type: Superiority; p = 0.204, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse Events were not collected.
Description: This was an observational study and not designed to assess adverse events; therefore, safety reporting was not applicable for this study.
Arm/Group | Crohn's Disease (Vedolizumab) | Crohn's Disease (Ustekinumab) | Ulcerative Colitis (Vedolizumab) | Ulcerative Colitis (Tofacitinib)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT04852666/Prot_SAP_000.pdf